CLINICAL TRIAL: NCT06232707
Title: A Phase 3, Randomized, Multicenter, Open-label Study to Evaluate the Efficacy and Safety of Alnuctamab Compared to Standard of Care Regimens in Participants With Relapsed or Refractory Multiple Myeloma (RRMM) - ALUMMINATE RRMM
Brief Title: A Study to Evaluate Efficacy and Safety of Alnuctamab Compared to Standard of Care Regimens in Participants With Relapsed or Refractory Multiple Myeloma (RRMM)
Acronym: ALUMMINATE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA058-1019; 2023-509472-42 (Registry Identifier: EU Trial Number); U1111-1281-8227 (Registry Identifier: WHO)
Record Dates: First submitted 2024-01-22; First posted 2024-01-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Multiple Myeloma
Keywords: Relapsed or Refractory Multiple Myeloma; BMS-986349; CC-93269; RRMM; Alnuctamab; CA058-1019; ALUMMINATE RRMM
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — pomalidomide; daratumumab; elotuzumab; carfilzomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Alnuctamab (Experimental)
  Interventions: Drug: Alnuctamab
- Arm B: Standard of Care Regimens (Active Comparator)
  Interventions: Drug: Pomalidomide; Drug: Daratumumab; Drug: Elotuzumab; Drug: Carfilzomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Alnuctamab — Specified dose on specified days
  Other Names: BMS-986349; CC-93269
  Arms: Arm A: Alnuctamab
Drug: Pomalidomide — Specified dose on specified days
  Other Names: POMALYST®; IMNOVID®; CC-4047; BMS-986379
  Arms: Arm B: Standard of Care Regimens
Drug: Daratumumab — Specified dose on specified days
  Other Names: DARZALEX®; DARZALEX; FASPRO®
  Arms: Arm B: Standard of Care Regimens
Drug: Elotuzumab — Specified dose on specified days
  Other Names: Empliciti®; BMS-901608
  Arms: Arm B: Standard of Care Regimens
Drug: Carfilzomib — Specified dose on specified days
  Other Names: KYPROLIS®
  Arms: Arm B: Standard of Care Regimens
Drug: Dexamethasone — Specified dose on specified days
  Arms: Arm B: Standard of Care Regimens

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of alnuctamab compared to standard of care regimens in participants with relapsed or refractory multiple myeloma (RRMM).

ELIGIBILITY:
Inclusion Criteria

* Participant is willing and able to adhere to the study visit schedule and other protocol requirements including bone marrow aspirations and/or biopsies and hospitalization during the first cycle.
* Documented diagnosis of multiple myeloma (MM), and must:.

  i) Received at least 1 but not more than 3 prior lines of anti-myeloma therapy.

ii) Received prior treatment with lenalidomide and an anti-CD38 monoclonal antibody (for at least 2 consecutive cycles).

iii) Achieved minimal response (MR) or better to at least 1 prior anti-myeloma therapy.

iv) Documented PD during or after their last anti-myeloma therapy or failure to achieve response.

* Must have measurable disease (as determined by central laboratory).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2 at the time of the screening.

Exclusion Criteria

* Active, uncontrolled, or suspected infection.
* Known current, or history of, central nervous system involvement of multiple myeloma.
* History or presence of clinically relevant CNS pathology.
* Received prior BCMA-targeted TCE or BCMA-targeted CAR-T therapy.
* Previously received allogeneic stem cell transplantation at any time or received autologous stem cell transplantation within 3 months of initiating study intervention.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-05-03 (Estimated); Primary Completion 2025-11-16 (Estimated); Study Completion 2030-09-21 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Up to 5 years

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 5 years
Overall response (OR) | Up to 5 years
Complete response (CR) or better | Up to 5 years
Very good partial response (VGPR) or better | Up to 5 years
Time to response (TTR) | Up to 5 years
Duration of response (DOR) | Up to 5 years
Time to progression (TTP) | Up to 5 years
Time to next treatment (TTNT) | Up to 5 years
Progression-free survival 2 (PFS2) | Up to 5 years
Restricted mean DOR (RMDOR) | Up to 5 years
Minimal residual disease (MRD) negativity rate | Up to 5 years
Incidence of adverse events (AEs) | Up to 5 years
Incidence of serious adverse events (SAEs) | Up to 5 years
Change from baseline in subscale scores of European organization for research and treatment of cancer - quality of life core 30 (EORTC QLQ-C30) | Up to 5 years
Change from baseline in subscale scores of European quality of life multiple myeloma module (EORTC QLQ-MY20) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (170):
- United States (22):
  - Local Institution - 0151, Birmingham, Alabama
  - Local Institution - 0088, Los Angeles, California
  - Local Institution - 0358, Stanford, California
  - Local Institution - 0355, New Haven, Connecticut
  - Local Institution - 0434, Washington D.C., District of Columbia
  - Local Institution - 0433, Wichita, Kansas
  - Local Institution - 0439, Saint Matthews, Kentucky
  - Local Institution - 0323, New Orleans, Louisiana
  - Local Institution - 0324, Baltimore, Maryland
  - Local Institution - 0441, Bethesda, Maryland
  - Local Institution - 0435, Billings, Montana
  - Local Institution - 0157, Hackensack, New Jersey
  - Local Institution - 0359, Summit, New Jersey
  - Local Institution - 0430, Lake Success, New York
  - Local Institution - 0396, New York, New York
  - Local Institution - 0306, Cincinnati, Ohio
  - Local Institution - 0199, Cleveland, Ohio
  - Local Institution - 0437, Pittsburgh, Pennsylvania
  - Local Institution - 0352, Providence, Rhode Island
  - Local Institution - 0420, Watertown, South Dakota
  - Local Institution - 0168, Dallas, Texas
  - Local Institution - 0405, Seattle, Washington
- Argentina (4):
  - Local Institution - 0001, La Plata, Buenos Aires
  - Local Institution - 0262, Pilar, Buenos Aires
  - Local Institution - 0222, San Juan Bautista, Buenos Aires
  - Local Institution - 0002, Buenos Aires, Buenos Aires F.D.
- Australia (8):
  - Local Institution - 0260, Liverpool, New South Wales
  - Local Institution - 0246, Macquarie University, New South Wales
  - Local Institution - 0022, Waratah, New South Wales
  - Local Institution - 0397, Brisbane, Queensland
  - Local Institution - 0021, Box Hill, Victoria
  - Local Institution - 0019, Clayton, Victoria
  - Local Institution - 0018, Melbourne, Victoria
  - Local Institution - 0003, Melbourne, Victoria
- Austria (4):
  - Local Institution - 0333, Sankt Pölten, Lower Austria
  - Local Institution - 0337, Innsbruck, Tyrol
  - Local Institution - 0334, Salzburg
  - Local Institution - 0332, Vienna
- Belgium (4):
  - Local Institution - 0284, Brasschaat, Antwerpen
  - Local Institution - 0280, Verviers, Liège
  - Local Institution - 0279, Yvoir, Namur
  - Local Institution - 0286, Leuven, Vlaams-Brabant
- Brazil (5):
  - Local Institution - 0274, Belo Horizonte, Minas Gerais
  - Local Institution - 0351, Natal, Rio Grande do Norte
  - Local Institution - 0369, São Paulo, São Paulo
  - Local Institution - 0291, Rio de Janeiro
  - Local Institution - 0211, São Paulo
- Canada (6):
  - Local Institution - 0417, Calgary, Alberta
  - Local Institution - 0423, Edmonton, Alberta
  - Local Institution - 0402, London, Ontario
  - Local Institution - 0395, Toronto, Ontario
  - Local Institution - 0031, Montreal, Quebec
  - Local Institution - 0098, Montreal, Quebec
- Chile (4):
  - Local Institution - 0027, Santiago, Metropolitana de Santiago
  - Local Institution - 0030, Santiago, Santiago Metropolitan
  - Local Institution - 0026, Santiago, Santiago Metropolitan
  - Local Institution - 0029, Santiago, Santiago Metropolitan
- China (30):
  - Local Institution - 0413, Beijing, Beijing Municipality
  - Local Institution - 0230, Beijing, Beijing Municipality
  - Local Institution - 0040, Beijing, Beijing Municipality
  - Local Institution - 0366, Changping, Beijing Municipality
  - Local Institution - 0057, Chongqing, Chongqing Municipality
  - Local Institution - 0066, Guangzhou, Guangdong
  - Local Institution - 0080, Guangzhou, Guangdong
  - Local Institution - 0226, Guangzhou, Guangdong
  - Local Institution - 0368, Shenzhen, Guangdong
  - Local Institution - 0365, Baoding, Hebei
  - Local Institution - 0082, Shijiazhuang, Hebei
  - Local Institution - 0041, Zhengzhou, Henan
  - Local Institution - 0075, Wuhan, Hubei
  - Local Institution - 0062, Changsha, Hunan
  - Local Institution - 0053, Changsha, Hunan
  - Local Institution - 0055, Nanjing, Jiangsu
  - Local Institution - 0067, Suzhou, Jiangsu
  - Local Institution - 0377, Xuzhou, Jiangsu
  - Local Institution - 0044, Shenyang, Liaoning
  - Local Institution - 0072, Xi'an, Shaanxi
  - Local Institution - 0077, Jinan, Shandong
  - Local Institution - 0083, Jinan, Shandong
  - Local Institution - 0273, Shanghai, Shanghai Municipality
  - Local Institution - 0421, Shanghai, Shanghai Municipality
  - Local Institution - 0245, Taiyuan, Shanxi
  - Local Institution - 0056, Tianjin, Tianjin Municipality
  - Local Institution - 0422, Tianjin, Tianjin Municipality
  - Local Institution - 0070, Hangzhou, Zhejiang
  - Local Institution - 0203, Hangzhou, Zhejiang
  - Local Institution - 0367, Qingdao
- Czechia (3):
  - Local Institution - 0013, Brno, Brno-město
  - Local Institution - 0247, Olomouc, Olomoucký kraj
  - Local Institution - 0012, Prague
- France (6):
  - Local Institution - 0118, Toulouse, Haute-Garonne
  - Local Institution - 0225, Montpellier, Languedoc-Roussillon
  - Local Institution - 0224, Vandœuvre-lès-Nancy, Lorraine
  - Local Institution - 0084, Lille, Nord
  - Local Institution - 0085, Nantes, Pays de la Loire Region
  - Local Institution - 0192, Pierre-Bénite, Rhône
- Germany (5):
  - Local Institution - 0331, Heidelberg, Baden-Wurttemberg
  - Local Institution - 0330, Tübingen, Baden-Wurttemberg
  - Local Institution - 0335, Dresden, Saxony
  - Local Institution - 0329, Leipzig, Saxony
  - Local Institution - 0339, Hamburg
- Greece (2):
  - Local Institution - 0004, Athens, Attikí
  - Local Institution - 0136, Chaïdári, Attikí
- Hungary (4):
  - Local Institution - 0103, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Local Institution - 0108, Szombathely, Vas County
  - Local Institution - 0104, Budapest
  - Local Institution - 0105, Budapest
- India (5):
  - Local Institution - 0370, Visakhapatnam, Andhra Pradesh
  - Local Institution - 0362, Gurugram, Haryana
  - Local Institution - 0403, Bangalore, Karnataka
  - Local Institution - 0399, Lucknow, Uttar Pradesh
  - Local Institution - 0398, Kolkata, West Bengal
- Ireland (4):
  - Local Institution - 0281, Cork
  - Local Institution - 0371, Dublin
  - Local Institution - 0285, Dublin
  - Local Institution - 0269, Limerick
- Italy (4):
  - Local Institution - 0096, Meldola, Emilia-Romagna
  - Local Institution - 0294, Legnano, Milano
  - Local Institution - 0265, Milan, Milano
  - Local Institution - 0410, Palermo, Sicily
- Japan (14):
  - Local Institution - 0409, Anjo, Aichi-ken
  - Local Institution - 0387, Nagoya, Aichi-ken
  - Local Institution - 0407, Kamogawa, Chiba
  - Local Institution - 0385, Kashiwa, Chiba
  - Local Institution - 0386, Isehara, Kanagawa
  - Local Institution - 0390, Ōsaka-sayama, Osaka
  - Local Institution - 0381, Shimotsuga, Tochigi
  - Local Institution - 0382, Koto, Tokyo
  - Local Institution - 0419, Aomori
  - Local Institution - 0383, Chiba
  - Local Institution - 0391, Kumamoto
  - Local Institution - 0389, Kyoto
  - Local Institution - 0388, Okayama
  - Local Institution - 0384, Tokyo
- Norway (3):
  - Local Institution - 0137, Løenskog, Akershus
  - Local Institution - 0115, Bergen, Hordaland
  - Local Institution - 0193, Oslo
- Portugal (3):
  - Local Institution - 0242, Lisbon, Lisbon District
  - Local Institution - 0415, Lisbon, Lisbon District
  - Local Institution - 0255, Lisbon
- Romania (3):
  - Local Institution - 0169, Bucharest, București
  - Local Institution - 0171, Brasov
  - Local Institution - 0414, Bucharest
- South Korea (6):
  - Local Institution - 0240, Seongnam, Kyǒnggi-do
  - Local Institution - 0221, Busan, Pusan-Kwangyǒkshi
  - Local Institution - 0036, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0239, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0034, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0035, Seoul, Seoul-teukbyeolsi [Seoul]
- Spain (7):
  - Local Institution - 0011, Badalona, Barcelona [Barcelona]
  - Local Institution - 0234, El Palmar, Murcia, Murcia, Región de
  - Local Institution - 0008, Pamplona, Navarre
  - Local Institution - 0202, Jerez de la Frontera
  - Local Institution - 0006, Salamanca
  - Local Institution - 0007, Santiago de Compostela
  - Local Institution - 0009, Valencia
- Sweden (2):
  - Local Institution - 0114, Borås, Västra Götalands Län [se-14]
  - Local Institution - 0111, Gothenburg, Västra Götalands Län [se-14]
- Switzerland (3):
  - Local Institution - 0336, Bern, Canton of Bern
  - Local Institution - 0411, Sankt Gallen, Canton of St. Gallen
  - Local Institution - 0338, Zurich
- Turkey (Türkiye) (4):
  - Local Institution - 0325, Stanbul, Istanbul
  - Local Institution - 0375, Ankara
  - Local Institution - 0188, Izmir
  - Local Institution - 0187, Kayseri
- United Kingdom (5):
  - Local Institution - 0349, Southampton, Hampshire
  - Local Institution - 0342, London, London, City of
  - Local Institution - 0350, Cardiff
  - Local Institution - 0344, Derby
  - Local Institution - 0343, Manchester

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome